CLINICAL TRIAL: NCT04913753
Title: Relevance of the Urine Bacterial Culture Performed Before Double J Ablation for Post-operative Urinary Tract Infection Prevention
Acronym: AblaJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR200086 - ABLAJ
Record Dates: First submitted 2021-05-19; First posted 2021-06-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Urinary Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No systematic CBEU (Experimental): Patients will not have bacterial culture performed before double J removal.
  Interventions: Procedure: No CBEU
- Systematic CBEU (Active Comparator): Patients will have a systematic urine culture performed before double J removal.
  Interventions: Procedure: CBEU

INTERVENTIONS:
Procedure: CBEU — Patients in the control group will have bacterial culture and double J removal will be performed as usual. .
  Arms: Systematic CBEU
Procedure: No CBEU — Patients in the experimental group will have bacterial culture and double J removal will be performed as usual. .
  Arms: No systematic CBEU

SUMMARY:
The value of cytobacteriological examination of urine (CBEU) before double J catheter removal has not been demonstrated. The aim of this study is to define the interest of this CBEU.

DETAILED DESCRIPTION:
Double J stents are ureteral catheters that allow urine to flow from the kidney without difficulty. These catheters protect the ureterovesical anastomosis of a renal transplant or reduce the postoperative oedema, for example after stone removal by ureteroscopy. These catheters are removed in an outpatient setting under local anaesthesia. Post ablation infections of double J catheters have been poorly studied but their incidence varied according to the populations and the definition used (10 to 54% for colonization, 1 to 10% for symptomatic infection). The national and international guidelines advocate a routine urine bacterial culture (UBC) before double J catheter removal as the procedure is in contact with urine; but there is no evidence of its interest. In case of positivity of this culture, it is recommended to delay the intervention or, what is more often chosen, to treat with antibiotic to cover the procedure. Investigators can thus ask 2 questions: is it rightful to withdraw a double J removal while the UBC is falsely negative and in case of a positive bacterial culture is there an increased risk of post-ablation infection?

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥ 18 years of age
* Scheduled to have a double J catheter ablation
* Participants covered by or entitled to social security
* Written informed consent obtained from the participant
* Ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Patients already receiving antibiotics other than urological reasons and transplanted patients
* Study interventions contraindications
* Pregnancy, breastfeeding
* Patient under tutorship or curators
* Deprivation of liberty

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Incidence of infection | 1 month post double J removal
  Incidence over a month period of post-ablation symptomatic urinary infection defined by the presence of symptoms validated by an adjudication committee (urine burning, fever, urgencies… associated to a significant bacteriuria) - each patient will be contacted by phone at month 1 (± 5 days) and will be asked to contact us in case of suspicion of urinary infection.

SECONDARY OUTCOMES:
Incidence of bacteriuria measured by CBEU | 1 month post double J removal
  Incidence of post-ablation bacteriuria (urosepsis and antibiotic use) in different groups of patients (reason of the stent, duration of the insertion, previous infection, immunodepression….) in the 1 month post-ablation period
Description of the resistance type of pre-operative distribution of bacteriuria by CBEU | 10 days to 4 days before double J removal
  Epidemiology of the resistance type of pre-operative bacteriuria
Description of the pre-operative distribution of bacteriuria by CBEU | 10 days to 4 days before double J removal
  Epidemiology of pre-operative bacteriuria
Description of the resistance type of post operative distribution of bacteriuria by CBEU | 1 month after double J removal
  Epidemiology of the resistance type of post-ablation bacteriuria
Description of the post operative distribution of bacteriuria by CBEU | 1 month after double J removal
  Epidemiology of post-ablation bacteriuria
Composition of microbiome by bacterial urinary analysis | 1 month post double J removal
  Comparison of the pre-operative urinary microbiome to the post-ablation urinary microbiome in patient with post-ablation infection.
Health-economic outcome | 1 month post double J removal
  Proportion of incremental costs-effects pairs that lies in the non-inferiority area, for various values of economic non-inferiority

CONTACTS AND LOCATIONS:
Locations (1):
- BRUYERE, Tours, France